CLINICAL TRIAL: NCT04677166
Title: Coupling Negative Pressure Wound Therapy With Instillation for Optimal Graft Take: Randomized Prospective Pilot Study
Brief Title: Coupling Negative Pressure Wound Therapy With Instillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At the American Society of Plastic Surgeons 2024 Meeting, an abstract was presented demonstrating substantial superiority of the technology employed in the experimental arm of this study versus the control.
Sponsor: Loma Linda University (Other)
Collaborators: Acelity (Other); KCI USA, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5200176
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Wound; Ulcer; Burns
MeSH Terms: conditions — Wounds and Injuries; Ulcer; Burns

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either the treatment group (negative pressure wound therapy coupled with instillation) or the control group (standard negative pressure wound therapy). Both groups will receive four days of intervention and outcomes will be measured at day four of negative pressure wound therapy and at thirty days post-operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NPWT with Instillation (Experimental): NPWT coupled with instillation will be employed via use of V.A.C. VeraFlo device. The protocol to be used is as follows:
  Instillation Solution: normal saline Dwell/Soak Time: 30 seconds Cycle Time: 4 hours Pressure: 125mmHg
  Interventions: Device: Negative pressure wound therapy coupled with instillation
- Standard NPWT (Active Comparator): Standard NPWT with use of V.A.C. Ulta device employed at 125mmHg continuous suction.
  Interventions: Device: Standard Negative Pressure Wound Therapy

INTERVENTIONS:
Device: Negative pressure wound therapy coupled with instillation — Use of V.A.C. VeraFlo to treat skin grafts with NPWT coupled with instillation.
  Arms: NPWT with Instillation
Device: Standard Negative Pressure Wound Therapy — standard negative pressure wound therapy via V.A.C. Ulta device at 125mmHg suction.
  Arms: Standard NPWT

SUMMARY:
The objective of this study is to compare standard negative pressure wound therapy with negative pressure wound therapy coupled with instillation for optimal skin graft take. Either the V.A.C ULTA NPWT or V.A.C. VeraFlo Therapy systems with normal saline will be applied intra-operatively to split-thickness skin grafts of upper and lower extremity wounds and kept in place for a duration of four days. Following completion of four days, the skin graft with be assessed for percentage of take/adherence and will be covered with simple gauze dressings as needed.

DETAILED DESCRIPTION:
Past studies have investigated the use of NPWT for post-operative skin graft treatment and shown superior outcomes regarding graft take and need for repeat grafting when compared with standard gauze dressing. However, to date, no study has compared standard NPWT to NPWT coupled with instillation for post-operative treatment of extremity skin grafts. This study is designed as a randomized, controlled pilot study to compare treatment standard NPWT with NPWT coupled with instillation on skin graft take.

Patients will be selected based on inclusion criteria and randomized to either the treatment (NPWT coupled with instillation) or the control group (standard NPWT). Depending on the group to which they are randomized to, patients will have standard NPWT or NPWT coupled with instillation applied intra-operatively after application of split thickness skin graft for treatment of extremity wound.

Patients randomized to control group will receive V.A.C Ulta NPWT at 125mmHg continuous pressure for duration of four days.

Patients randomized to treatment group will receive V.A.C VeraFlo therapy. Protocol will consist of the following:

* Instillation solution: normal saline
* Dwell/soak time: 30 seconds
* Cycle Time: 4 hours
* Pressure: 125mmHg

The devices will be kept in place for four days, at which point, the wound vacs will be removed and the percentage of skin graft take will be evaluated with use of photometric analysis. The skin grafts will be subsequently dressed with gauze as appropriate. Patients will be followed up in clinic to assess outcome of skin graft take.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been offered split-thickness skin graft for treatment of an extremity wound.

Exclusion Criteria:

* Abnormal healing (diagnosed with connective tissue disorder)
* Uncontrolled diabetes mellitus (HgbA1c >9)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Skin Graft Take at Four Days Post-Operative | 4 days from intervention
  percentage of skin graft take at time of wound vac take down (4 days post-op)

SECONDARY OUTCOMES:
Percentage of Skin Graft Take at Thirty Days Post-Operative | 30 days from intervention
  percentage of skin graft take at follow up clinic appointment

CONTACTS AND LOCATIONS:
Overall Officials: Subhas W Gupta, MD, PhD, Principal Investigator — Loma Linda
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yin Y, Zhang R, Li S, Guo J, Hou Z, Zhang Y. Negative-pressure therapy versus conventional therapy on split-thickness skin graft: A systematic review and meta-analysis. Int J Surg. 2018 Feb;50:43-48. doi: 10.1016/j.ijsu.2017.12.020. Epub 2017 Dec 29. PMID 29292216
- [Background] Nguyen TQ, Franczyk M, Lee JC, Greives MR, O'Connor A, Gottlieb LJ. Prospective randomized controlled trial comparing two methods of securing skin grafts using negative pressure wound therapy: vacuum-assisted closure and gauze suction. J Burn Care Res. 2015 Mar-Apr;36(2):324-8. doi: 10.1097/BCR.0000000000000089. PMID 25162948